CLINICAL TRIAL: NCT03000387
Title: Personalized Dosing of Nicotine Replacement for Smoking Cessation: An Effectiveness Randomized Placebo-controlled Trial
Brief Title: Personalized Dosing of Nicotine Replacement (NRT to Effect)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Laurie Zawertailo, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 039/2015
Record Dates: First submitted 2016-11-17; First posted 2016-12-22 (Estimated); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Tobacco Use Disorder; Nicotine Dependence
Keywords: Nicotine Replacement Therapy; Smoking Cessation; Randomized Clinical Trial; Nicotine Patch; Abstinence; Placebo; Double blind
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Condition (Experimental): Participants unable to quit smoking after 2 weeks of treatment with 21mg nicotine patch will get 21mg nicotine patches plus additional active nicotine patches until achieving 7 consecutive days of abstinence over the next 5 weeks; maximum daily patch dose, 84mg/day
  Interventions: Drug: Nicotine Patch
- Placebo Condition (Placebo Comparator): Participant unable to quit smoking after 2 weeks of treatment with 21mg nicotine patch will get 21mg nicotine patches plus placebo patches until 7 consecutive days of abstinence over the next 5 weeks; Maximum daily patch dose, 21mg active nicotine patch plus 3 placebo 21mg patches.
  Interventions: Drug: Nicotine Patch; Drug: Placebos
- Quit condition (Active Comparator): Participants able to quit for 7 consecutive days during the first 2 weeks of treatment with 21mg nicotine patch will continue open label 21mg active nicotine patches for the remaining 10 weeks.
  Interventions: Drug: Nicotine Patch

INTERVENTIONS:
Drug: Nicotine Patch — Active nicotine patch of 21 mg, 14 mg and 7 mg
  Other Names: Nicoderm
Drug: Placebos — Matching placebo patches of 21 mg, 14 mg and 7 mg
  Other Names: Placebo patch
  Arms: Placebo Condition

SUMMARY:
Medications for smoking cessation are currently only effective in helping a minority of smokers quit. Drug development is slow and expensive, so there is much interest in optimizing the effectiveness of existing treatments and medications. Current standard doses of nicotine replacement therapy (NRT) are not effective for many smokers and in many cases provide less nicotine compared to when a smoker is smoking their usual number of cigarettes. The proposed study will test if a personalized dose of nicotine patch (up to 84mg) will improve quitting success in those who do not respond to a standard dose of NRT (21mg).

DETAILED DESCRIPTION:
A total of 500 smokers will be enrolled from two smoking cessation clinics to participate in this study. After 2 weeks of usual treatment with 21mg patch, participants who fail to quit smoking will be randomized to receive either escalating doses of active nicotine patches, or placebo patches, for 10 weeks. Those who stop smoking during the first 2 weeks of usual treatment will continue with 21mg patch treatment for 10 weeks as an additional comparison group. In addition to the medication, participants in all groups will receive brief behavioral counselling. Subjects will return to the clinic at weeks 26 and 52 to assess whether or not they are still abstinent from smoking and self-reports of non-smoking will be confirmed using a urine test for nicotine by-product (cotinine) levels. Exhaled carbon monoxide (CO) will be recorded as an additional measure. Study follow-up visits can be conducted virtually if needed.

The goal of the proposed study is to optimize the current gold standard smoking cessation treatment (nicotine patch plus brief counseling) in order to further increase quit rates. Evidence supporting the effectiveness of personalized doses of NRT could change current practice in a wide variety of healthcare settings. Given the strong link between smoking and cancer, and evidence that quitting smoking at any age diminishes this risk, even small increases in absolute quit rates can have a substantial population-level impact on reducing the incidence of smoking-related cancers, reducing mortality rates and associated healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

1. Daily tobacco smoker of ≥10 cigarettes per day
2. Aged 18 to 75 years old
3. Interested in using tNRT as the only smoking cessation aid
4. Intending to quit smoking within the next 30 days

Exclusion Criteria:

1. At least weekly use of tobacco products other than cigarettes and not willing to stop for the duration of the study
2. Breast feeding, pregnancy or not using a reliable form of birth control
3. Any generalized skin disorders precluding the use of the patch
4. Any life threatening arrhythmias or severe/worsening angina pectoris or within two weeks of experiencing a myocardial infarction or cerebral vascular accident
5. Currently using or has used NRT or other smoking cessation pharmacotherapy within the past two weeks
6. Any known hypersensitivity or allergies to any of the components comprising the nicotine patch
7. Current active substance dependence (excluding caffeine) which would compromise study compliance
8. Current unstable psychiatric condition which would compromise study compliance
9. Diagnosis of terminal illness
10. Current regular use of e-cigarettes or other vaping devices containing nicotine and not willing to stop for the duration of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Short term continuous abstinence | weeks 9 to 12
  YES, If self-reported 4 weeks of abstinence without a single puff of a cigarette or any other tobacco product. Else, NO.

SECONDARY OUTCOMES:
Long term continuous abstinence | weeks 9-26
  YES, if self-reported abstinence without a single puff of cigarette and urine cotinine less than 200ng/ml. Else, NO.
Long term continuous abstinence | weeks 9-52
  YES, if, self-reported abstinence without a single puff of cigarette and urine cotinine less than 200ng/ml. Else, NO.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Zawertailo, PhD, Principal Investigator — Centre for Addiction and Mental Health; Peter Selby, MBBS, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995
- [Derived] Zawertailo L, Hendershot CS, Tyndale RF, Le Foll B, Samokhvalov AV, Thorpe KE, Pipe A, Reid RD, Selby P. Personalized dosing of nicotine replacement therapy versus standard dosing for the treatment of individuals with tobacco dependence: study protocol for a randomized placebo-controlled trial. Trials. 2020 Jun 29;21(1):592. doi: 10.1186/s13063-020-04532-7. PMID 32600406